CLINICAL TRIAL: NCT04156152
Title: Effectiveness of the Use of Desensitizing Dentifrices Based on Nanocrystals of Hydroxyapatite / 5% Potassium Nitrate / 1450ppm Sodium Monofluorophosphate and Potassium Nitrate 5% / 1426ppm Sodium Floride in the Treatment of Dentine Hypersensitivity. Test Randomized Clinical
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Florencia Pacheco (Unknown)
Responsible Party: Principal Investigator, Francesca Lo Presti Arellano, Alumn Periodonthics UDD, Universidad del Desarrollo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2019-09-26; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Hypersensitivity Dentin
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be conducted to compare the clinical efficacy in reducing dentinal hypersensitivity in patients treated with dentifrices based on hydroxyapatite / 5% potassium nitrate / sodium monofluorophosphate 1450 ppm and 5% potassium nitrate / 1426ppm sodium fluoride, during an evaluation period of 8 weeks.
Who Masked: Participant, Care Provider
Masking Description: The masking will be done by concealing the two main faces of the dentifrice container with a white adhesive and this will be delivered in sealed packages, all of the same color and shape.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Grupo I (Active Comparator): 16 patients
  Interventions: Other: DEENSIBILIZING TOOTHPASTE BASED ON NANOCRISTALS OF HYDROXIAPATITA / 5% POTASSIC NITRATE / SODIUM MONOFluORPHOSPHATE 1450 PARTS PER MILLION
- Grupo II (Active Comparator): 16 patients
  Interventions: Other: 5% POTASSIC NITRATE / SODIUM FLUORIDE 1426 PARTS PER MILLION TOOTHPASTE

INTERVENTIONS:
Other: DEENSIBILIZING TOOTHPASTE BASED ON NANOCRISTALS OF HYDROXIAPATITA / 5% POTASSIC NITRATE / SODIUM MONOFluORPHOSPHATE 1450 PARTS PER MILLION — The toothpastes will be delivered by the researchers and will be applied with a manual toothbrush, with soft bristles and straight handle, by the patient.The 2nd, 3rd, 4th session (2nd, 4th, 6th week of follow-up) will be the application of tests and reinforcement of oral hygiene instruction. In the 5th session (8th week of follow-up) the pastes will be requested to verify compliance.
  Arms: Grupo I
Other: 5% POTASSIC NITRATE / SODIUM FLUORIDE 1426 PARTS PER MILLION TOOTHPASTE — The toothpastes will be delivered by the researchers and will be applied with a manual toothbrush, with soft bristles and straight handle, by the patient.The 2nd, 3rd, 4th session (2nd, 4th, 6th week of follow-up) will be the application of tests and reinforcement of oral hygiene instruction. In the 5th session (8th week of follow-up) the pastes will be requested to verify compliance.
  Arms: Grupo II

SUMMARY:
Background: Currently, periodontal treatment, both surgical and non-surgical, leaves sequelae in the vast majority of patients, dentine hypersensitivity (HSD) is one of the most important. For this reason, it is necessary to correctly diagnose this condition, to achieve a correct treatment of it. HSD is a condition frequently, which has been described as acute, provoked pain, which is not attributable to any other dental pathology. Its current prevalence is unknown, but it occurs in most patients after their periodontal treatment, and also in healthy patients.

Course objective: To compare the clinical efficacy in reducing dentinal hypersensitivity in patients treated with dentifrices based on hydroxyapatite / 5% potassium nitrate / sodium monofluorophosphate 1450ppm and 5% potassium nitrate / 1426ppm sodium fluoride, during a period of evaluation of 8 weeks Materials and methods: A randomized clinical trial will be conducted. Inclusion criteria will be: patients ≥ 18 years, dentinal hypersensitivity in at least one tooth (incisors, canines, premolars) of analogous visual scale ≥4, healthy patients and patients with pathologies, controlled, absence of pathologies that contraindicate participation in the study. Exclusion criteria will include: teeth with extensive or defective fillings, tooth decay and pulpitis, dental crack, unit fixed prosthesis and plural fixed prosthesis, pregnant patients, regular anti-inflammatory treatment, allergy to any of the components of the study, hypersensitivity treatment Recent dentistry Patients will be assigned to two groups. The experimental group (n = 16) will be delivered with hydroxyapatite nanocrystals (VITIS® sensitive) and the control group (n = 16) will be given a paste with 5% potassium nitrate (Sensodyne True White), and after performing an instruction for use on the first visit, four subsequent visits will be made at 2, 4, 6 and 8 weeks after the initial visit. At each visit the hard and soft tissue exam will be performed; and also cold, heat, evaporative and electrical tests will be carried out on the teeth that will be included in the study. The tests will be performed by two previously calibrated researchers, and then the results will be entered into a computer program to perform the effectiveness calculations.

Expected results: The results of the present study would demonstrate that there is a general decrease in dentinal hypersensitivity in both groups, during the 8-week study period, presenting a significantly greater improvement in dentin hypersensitivity in either of the two control groups.

Keywords: Dentine hypersensitivity, desensitizing paste, hydroxyapatite, potassium nitrate.

DETAILED DESCRIPTION:
Currently, periodontal treatment, both surgical and non-surgical, leaves sequelae in the vast majority of patients. The loss of clinical insertion level could be an early indicator or a possible risk factor for dentine hypersensitivity (HSD) (15). Therefore, it is necessary to correctly diagnose this condition, to achieve a correct treatment of it, which can be performed both in the clinic and at home.

HSD is a condition frequently present in individuals, leading them to seek help from a dentist. It has been described as an acute, provoked pain, which is not attributable to any other dental pathology. Its current prevalence is unknown, but it occurs in most patients after their periodontal treatment, and also in healthy patients. (12) To determine the diagnosis and treatment of HSD, it is necessary to deepen the history, the assessment of the patient's pain through a self-assessment system such as the visual analogue scale (VAS), the differentiation between other pathologies using different tools and clinical interpretation, since that the ongoing processes that determine and maintain the opening and permeability of dentinal tubules are still under discussion. Multiple therapeutic modalities are used to manage HSD according to the intensity of pain and patient education, such as the use of remineralizing, desensitizing, blocking, analgesic dentifrices to restorative dentistry therapies, mucogingival surgeries, among others (14).

The research question of this study is: Is the application of a toothpaste based on hydroxyapatite / 5% potassium nitrate / sodium monofluorophosphate 1450ppm nano-crystals more effective compared to the application of a 5% potassium nitrate / fluoride toothpaste Sodium 1426ppm in the treatment of HSD? The general objective is to compare the clinical efficacy in reducing HSD in patients treated with dentifrices based on nano crystals of hydroxyapatite / 5% potassium nitrate / sodium monofluorophosphate 1450ppm and potassium nitrate 5% / sodium fluoride 1426ppm, during an evaluation period 8 weeks The importance of this study lies in the lack of information and quality studies that really assess the effectiveness of the various types of desensitizing toothpastes, so as to be clear about the most effective dentifrices and direct the dentist in the treatment of HSD

ELIGIBILITY:
The inclusion criteria that will be used for patient eligibility will be: Patients between 18 and 80 years old, HSD in at least two teeth (incisors, premolars, canines) VAS ≥4 and absence of pathologies that contraindicate participation in the study.

The exclusion criteria that will be addressed will be: Teeth with extensive or defective fillings, tooth decay and pulpitis, dental crack, unit fixed prosthesis and plural fixed prosthesis, pregnant patients, regular treatment with anti-inflammatories, allergy to any of the components of the study and / or recent dentin hypersensitivity treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-04-10 (Estimated); Primary Completion 2020-07-10 (Estimated); Study Completion 2020-08-21 (Estimated)

PRIMARY OUTCOMES:
Dentinal Hypersensitivity | 3 months
  The cold test will be carried out, through the application of TFE tetrafluoroethane.
Dentinal Hypersensitivity | 3 months
  The heat test will be carried out, by applying a hot gutta-percha bar (120-140 ° C)
Dentinal Hypersensitivity | 3 months
  The electrical test will be carried out, through the application of a vitalometer.
Dentinal Hipersensitivity | 3 months
  The evaporative test will be carried out, after relative isolation with the triple syringe of air

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langenbach F, Naujoks C, Smeets R, Berr K, Depprich R, Kubler N, Handschel J. Scaffold-free microtissues: differences from monolayer cultures and their potential in bone tissue engineering. Clin Oral Investig. 2013 Jan;17(1):9-17. doi: 10.1007/s00784-012-0763-8. Epub 2012 Jun 14. PMID 22695872
- [Background] Splieth CH, Tachou A. Epidemiology of dentin hypersensitivity. Clin Oral Investig. 2013 Mar;17 Suppl 1(Suppl 1):S3-8. doi: 10.1007/s00784-012-0889-8. Epub 2012 Dec 7. PMID 23224064
- [Background] Uraz A, Erol-Simsek O, Pehlivan S, Suludere Z, Bal B. The efficacy of 8% Arginine-CaCO(3) applications on dentine hypersensitivity following periodontal therapy: a clinical and scanning electron microscopic study. Med Oral Patol Oral Cir Bucal. 2013 Mar 1;18(2):e298-305. doi: 10.4317/medoral.17990. PMID 23229241
- [Background] Matis BA, Cochran MA, Eckert GJ, Matis JI. In vivo study of two carbamide peroxide gels with different desensitizing agents. Oper Dent. 2007 Nov-Dec;32(6):549-55. doi: 10.2341/07-10. PMID 18051004
- [Background] Gandolfi MG, Silvia F, H PD, Gasparotto G, Carlo P. Calcium silicate coating derived from Portland cement as treatment for hypersensitive dentine. J Dent. 2008 Aug;36(8):565-78. doi: 10.1016/j.jdent.2008.03.012. Epub 2008 Jun 6. PMID 18538913
- [Background] Cunha-Cruz J, Wataha JC, Heaton LJ, Rothen M, Sobieraj M, Scott J, Berg J; Northwest Practice-based Research Collaborative in Evidence-based DENTistry. The prevalence of dentin hypersensitivity in general dental practices in the northwest United States. J Am Dent Assoc. 2013 Mar;144(3):288-96. doi: 10.14219/jada.archive.2013.0116. PMID 23449905
- [Background] Kihn PW, Barnes DM, Romberg E, Peterson K. A clinical evaluation of 10 percent vs. 15 percent carbamide peroxide tooth-whitening agents. J Am Dent Assoc. 2000 Oct;131(10):1478-84. doi: 10.14219/jada.archive.2000.0061. PMID 11042989
- [Background] Haywood VB. Treating sensitivity during tooth whitening. Compend Contin Educ Dent. 2005 Sep;26(9 Suppl 3):11-20. PMID 17039676